CLINICAL TRIAL: NCT04284072
Title: A Multicenter Study to Examine Clinical Scenarios for Long-term Monitoring of Epileptic Seizures With a Wearable Biopotential Technology
Brief Title: Clinical Scenarios for Long-term Monitoring of Epileptic Seizures With a Wearable Biopotential Technology
Acronym: SeizeIT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Freiburg University (Unknown); King's College London (Other); Oxford University Hospitals NHS Trust (Other); University of Coimbra (Other); Karolinska Institutet (Other); RWTH Aachen University (Other); UCB Pharma (Industry); Byteflies (Industry); Helpilepsy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: S63631
Record Dates: First submitted 2020-02-17; First posted 2020-02-25 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-05

CONDITIONS: Epilepsy
Keywords: Seizure detection; Wearable; Epilepsy; Seizure; Sensor Dot
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Single arm study with a device intervention for epileptic seizure monitoring in subjects with refractory focal impaired awareness, tonic-clonic, and/or typical absence seizures.
  Interventions: Device: Sensor Dot

INTERVENTIONS:
Device: Sensor Dot — Multimodal (EEG, ECG, EMG and motion) seizure monitoring with Sensor Dot to complement EMU-based video-EEG monitoring (EMU Phase), and optional home-based seizure diary logging (Home Phase).

SUMMARY:
Clinically validate a biopotential and motion recording wearable device (Byteflies Sensor Dot) for detection of epileptic seizures in the epilepsy monitoring unit (EMU) and at home.

DETAILED DESCRIPTION:
Subjects with refractory epilepsy who are admitted to the Epilepsy Monitoring Unit (EMU) for clinically-indicated long-term video-EEG assessment will be simultaneously monitored with Sensor Dots to record electroencephalographic (EEG), electrocardiographic (ECG), electromyographic (EMG), and motion signals.

A subset of subjects will continue using Sensor Dot devices at home (Home Phase) after completing the EMU Phase.

The data recorded by Sensor Dots will be used to: 1) annotate epileptic seizures, which will be compared to the annotations made as part of routine EMU monitoring and seizure diaries kept at home, and 2) to develop seizure detection algorithms. The data collected as part of this study will not be used to influence clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (4+ years old) with refractory epilepsy who are admitted to the hospital for clinically-indicated long-term video-EEG assessment or presurgical evaluation, and a high likelihood of experiencing seizures during the EMU Phase
* For subjects continuing into the Home Phase: successful recording of their habitual seizures with Sensor Dot during the EMU Phase
* For subjects continuing into the Home Phase: the ability to keep an e-diary

Exclusion Criteria:

* Known allergies to any of the biopotential electrodes or adhesives used as part of the study protocol
* Having an implanted device, such as (but not limited to) a pacemaker, cardioverter defibrillator (ICD), and/or neural stimulation device because Sensor Dot contains magnets that could interfere with the operation of these devices
* Women who are pregnant

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison of typical absence seizure annotations derived from Sensor Dot data collected during the EMU Phase against annotations derived from video-EEG equipment during wakefulness | up to two weeks
  F1-score as determined by expert reviewers
Comparison of typical absence seizure annotations derived from Sensor Dot data collected during the EMU Phase against annotations derived from video-EEG equipment during sleep | up to two weeks
  F1-score as determined by expert reviewers
Comparison of focal impaired awareness seizure annotations derived from Sensor Dot data collected during the EMU Phase against annotations derived from video-EEG equipment during wakefulness | up to two weeks
  F1-score as determined by expert reviewers
Comparison of focal impaired awareness seizure annotations derived from Sensor Dot data collected during the EMU Phase against annotations derived from video-EEG equipment during sleep | up to two weeks
  F1-score as determined by expert reviewers
Comparison of tonic-clonic seizure annotations derived from Sensor Dot data collected during the EMU Phase against annotations derived from video-EEG equipment during wakefulness | up to two weeks
  F1-score as determined by expert reviewers
Comparison of tonic-clonic seizure annotations derived from Sensor Dot data collected during the EMU Phase against annotations derived from video-EEG equipment during sleep | up to two weeks
  F1-score as determined by expert reviewers

SECONDARY OUTCOMES:
Sensor Dot usability | up to two weeks
  We will assess the usability of the device as perceived by users (patients and healthcare personnel) via surveys
To assess seizure duration | up to two weeks
  From the Sensor Dot data, we will be able to assess seizure duration
To assess the usability of the seizure e-diary | up to two weeks
  We will asses usability of the electronic seizure diary
To evaluate the accuracy of automated seizure detection algorithms | 2 years
  We will use the collected data and seizure annotations to develop algorithms to automatically detect epileptic seizures. We plan to evaluate how accurate these new automated seizure detection algorithms are.
Comparison of seizure annotations derived from Sensor Dot data collected during the Home Phase against seizure diary annotations | up to 2 weeks
  Accuracy as determined by expert reviewers
Sensor Dot Performance | up to 2 weeks
  We will assess the technical performance of the device by comparing the actual length of recorded data against the expected recording length, and what percentage of the data is high quality enough to make seizure annotations.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Paesschen, MD, PhD, Principal Investigator — UZ Leuven and KU Leuven
Locations (7):
- University Hospitals Leuven, department of Neurology, Leuven, Belgium
- Germany (2):
  - Department of Epileptology and Neurology, Aachen
  - Epilepsy Center, University Medical Center, Freiburg University, Freiburg im Breisgau
- Division of Neurology, Coimbra University Hospital, Coimbra, Portugal
- Department of Clinical Neuroscience, Karolinska Institute, Stockholm, Sweden
- United Kingdom (2):
  - Division of Neuroscience, King's College London, London
  - Nuffield Department of Clinical Neurosciences, Oxford University Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the individual biosignals (EEG, EMG, ECG and movement) and 24-channel seizure-annotated EEG data, de-identified demographic and epilepsy-related data two years after the finish of the study (1-1-2024) upon request to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol
Time Frame: Data will be shared from 1-1-2024. We do not foresee an end-date.
Access Criteria: Data will be made available upon request to researchers who provide a methodologically sound proposal. Proposals should be directed to Wim.vanpaesschen@uzleuven.be

REFERENCES:
- [Background] Fisher RS, Acevedo C, Arzimanoglou A, Bogacz A, Cross JH, Elger CE, Engel J Jr, Forsgren L, French JA, Glynn M, Hesdorffer DC, Lee BI, Mathern GW, Moshe SL, Perucca E, Scheffer IE, Tomson T, Watanabe M, Wiebe S. ILAE official report: a practical clinical definition of epilepsy. Epilepsia. 2014 Apr;55(4):475-82. doi: 10.1111/epi.12550. Epub 2014 Apr 14. PMID 24730690
- [Background] Sander JW. The epidemiology of epilepsy revisited. Curr Opin Neurol. 2003 Apr;16(2):165-70. doi: 10.1097/01.wco.0000063766.15877.8e. PMID 12644744
- [Background] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Background] Elger CE, Hoppe C. Diagnostic challenges in epilepsy: seizure under-reporting and seizure detection. Lancet Neurol. 2018 Mar;17(3):279-288. doi: 10.1016/S1474-4422(18)30038-3. PMID 29452687
- [Background] Hoppe C, Poepel A, Elger CE. Epilepsy: accuracy of patient seizure counts. Arch Neurol. 2007 Nov;64(11):1595-9. doi: 10.1001/archneur.64.11.1595. PMID 17998441
- [Background] Kurada AV, Srinivasan T, Hammond S, Ulate-Campos A, Bidwell J. Seizure detection devices for use in antiseizure medication clinical trials: A systematic review. Seizure. 2019 Mar;66:61-69. doi: 10.1016/j.seizure.2019.02.007. Epub 2019 Feb 13. PMID 30802844
- [Background] Bidwell J, Khuwatsamrit T, Askew B, Ehrenberg JA, Helmers S. Seizure reporting technologies for epilepsy treatment: A review of clinical information needs and supporting technologies. Seizure. 2015 Nov;32:109-17. doi: 10.1016/j.seizure.2015.09.006. Epub 2015 Sep 18. PMID 26552573
- [Background] Beniczky S, Ryvlin P. Standards for testing and clinical validation of seizure detection devices. Epilepsia. 2018 Jun;59 Suppl 1:9-13. doi: 10.1111/epi.14049. PMID 29873827
- [Background] Szabo CA, Morgan LC, Karkar KM, Leary LD, Lie OV, Girouard M, Cavazos JE. Electromyography-based seizure detector: Preliminary results comparing a generalized tonic-clonic seizure detection algorithm to video-EEG recordings. Epilepsia. 2015 Sep;56(9):1432-7. doi: 10.1111/epi.13083. Epub 2015 Jul 20. PMID 26190150
- [Background] Beniczky S, Conradsen I, Wolf P. Detection of convulsive seizures using surface electromyography. Epilepsia. 2018 Jun;59 Suppl 1:23-29. doi: 10.1111/epi.14048. PMID 29873829
- [Background] Beniczky S, Polster T, Kjaer TW, Hjalgrim H. Detection of generalized tonic-clonic seizures by a wireless wrist accelerometer: a prospective, multicenter study. Epilepsia. 2013 Apr;54(4):e58-61. doi: 10.1111/epi.12120. Epub 2013 Feb 8. PMID 23398578
- [Background] Kjaer TW, Sorensen HBD, Groenborg S, Pedersen CR, Duun-Henriksen J. Detection of Paroxysms in Long-Term, Single-Channel EEG-Monitoring of Patients with Typical Absence Seizures. IEEE J Transl Eng Health Med. 2017 Jan 9;5:2000108. doi: 10.1109/JTEHM.2017.2649491. eCollection 2017. PMID 29018634
- [Background] Zibrandtsen IC, Kidmose P, Christensen CB, Kjaer TW. Ear-EEG detects ictal and interictal abnormalities in focal and generalized epilepsy - A comparison with scalp EEG monitoring. Clin Neurophysiol. 2017 Dec;128(12):2454-2461. doi: 10.1016/j.clinph.2017.09.115. Epub 2017 Oct 12. PMID 29096220
- [Background] Gu Y, Cleeren E, Dan J, Claes K, Van Paesschen W, Van Huffel S, Hunyadi B. Comparison between Scalp EEG and Behind-the-Ear EEG for Development of a Wearable Seizure Detection System for Patients with Focal Epilepsy. Sensors (Basel). 2017 Dec 23;18(1):29. doi: 10.3390/s18010029. PMID 29295522
- [Background] Dan J, Weckhuysen D, Cleeren E, Van Paesschen W, Vandendriessche B. Technical validation of Sensor Dot: a wearable for ambulatory monitoring of epileptic seizures. 2nd International Congress on mobile devices and seizure detection in epilepsy; Lausanne, Switzerland, 2019.
- [Background] Seeck M, Koessler L, Bast T, Leijten F, Michel C, Baumgartner C, He B, Beniczky S. The standardized EEG electrode array of the IFCN. Clin Neurophysiol. 2017 Oct;128(10):2070-2077. doi: 10.1016/j.clinph.2017.06.254. Epub 2017 Jul 17. PMID 28778476
- [Derived] Macea J, Heremans ERM, Proost R, De Vos M, Van Paesschen W. Automated Sleep Staging in Epilepsy Using Deep Learning on Standard Electroencephalogram and Wearable Data. J Sleep Res. 2025 Oct;34(5):e70061. doi: 10.1111/jsr.70061. Epub 2025 Apr 3. PMID 40176726
- See also: EIT Health website referring to our SeizeIT2 project — https://www.eithealth.eu/seizeit2